CLINICAL TRIAL: NCT02955862
Title: Vietnam Cryptococcal Retention in Care Study (CRICS) Federal Financial Report From June 2015 to June 2016
Brief Title: Vietnam Cryptococcal Retention in Care Study (CRICS) Federal Financial Report
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Hospital for Tropical Diseases, Hanoi, Vietnam (Other Government)
Responsible Party: Principal Investigator, Vu Quoc Dat, Lead Coordinator, National Hospital for Tropical Diseases, Hanoi, Vietnam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 3U01GH000758-02S1 (NIH)
Record Dates: First submitted 2016-10-28; First posted 2016-11-04 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Cryptococcal Meningitis
Keywords: Cryptococcal antigenemia; Cryptococcal meningitis; HIV/AIDS
MeSH Terms: conditions — Meningitis, Cryptococcal; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Assigned Interventions Antifungals Patients with symptoms (Other): Patients with symptoms of CNS disease will be treated according to Vietnam national guidelines for HIV/AIDS management.
  For CrAg-positive patients, the initial dosage of fluconazole will be 900 mg taken each day for 2 weeks. This will be followed by fluconazole 450 mg orally each day for 8 weeks. Finally, maintenance treatment with fluconazole 200mg orally each (2 tablets of 100 mg procured especially for the study) day will continue until CD4 >200 cells/µL for at least 6 months.
  Interventions: Other: Vietnam Cryptococcal Retention in Care Study (CRICS)

INTERVENTIONS:
Other: Vietnam Cryptococcal Retention in Care Study (CRICS) — Drug: Fluconazole HIV-infected patients with CD4 ≤100 cells/μL who present for HIV care at outpatient clinics (OPCs) in Vietnam where CrAg screening is offered will be recruited into the study. Study participants will be screened for cryptococcal antigen using the Lateral Flow Assay (LFA). Those who are CrAg-positive, but have no features of central nervous system (CNS) disease, will be treated with high-dose fluconazole.
  Other Names:
  • Fluconazole

SUMMARY:
CRICS financial report for the first budget year of the study

DETAILED DESCRIPTION:
Vietnam Cryptococcal Retention in Care Study (CRICS) federal financial report for the first budget year of the study

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Confirmed HIV infection using National Testing Algorithm
* CD4 ≤100 cells/μL
* Able to provide written informed consent

Exclusion Criteria:

* History of prior CM
* Receipt of systemic antifungal medication for more than 4 consecutive weeks within the past 6 months
* Currently taking ART or history of ART for more than 4 weeks within the past year
* Known to be currently pregnant or planning to become pregnant during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1177 (Actual)
Dates: Start 2015-06; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who have advanced HIV disease (CD4 <100) | 12 months
Prevalence of CrAg-positivity among HIV patients with advanced disease | 12 months
The proportion of patients who have no new opportunistic infections at 12 months | 12 months
Mortality rate among HIV patients with advanced disease | 12 months

SECONDARY OUTCOMES:
The proportion of patients with advanced HIV disease who retain in HIV care at 6 months and 12 months | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen V Kinh, Dr, Principal Investigator — NHTD
Locations (1):
- National hospital for tropical diseases, Ham Zong, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dat VQ, Lyss S, Dung NTH, Hung LM, Pals SL, Anh HTV, Kinh NV, Bateganya M. Prevalence of Advanced HIV Disease, Cryptococcal Antigenemia, and Suboptimal Clinical Outcomes Among Those Enrolled in Care in Vietnam. J Acquir Immune Defic Syndr. 2021 Dec 15;88(5):487-496. doi: 10.1097/QAI.0000000000002786. PMID 34446679